CLINICAL TRIAL: NCT00670436
Title: The Paclitaxel-Eluting PTCA-Balloon Catheter in Coronary Artery Disease to Treat Chronic Total Occlusions
Brief Title: The Paclitaxel-Eluting Percutaneous Transluminal Coronary Angioplasty (PTCA) - Balloon Catheter in Coronary Artery Disease to Treat Chronic Total Occlusions
Acronym: PEPCAD-CTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Principal Investigator, Jochen Wohrle, Prof. Dr. Jochen Wöhrle, University of Ulm
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPCAD-CTO V 2.3
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion; Native Coronary Artery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 1 (Active Comparator): paclitaxel eluting PTCA balloon (SeQuent please) after bare-metal stenting of a chronic total occlusion in a native coronary artery
  Interventions: Device: paclitaxel eluting PTCA balloon catheter (SeQuent Please)
- A2 (Active Comparator): historical population of patients with a chronic total occlusion in a native coronary artery treated with the paclitaxel eluting Taxus stent (Boston Scientific)
  Interventions: Device: paclitaxel eluting Taxus stent (Boston Scientific)

INTERVENTIONS:
Device: paclitaxel eluting PTCA balloon catheter (SeQuent Please) — paclitaxel eluting PTCA balloon catheter after bare-metal stenting of chronic total occlusion in a native coronary artery
  Other Names: SeQuent Please; paclitaxel eluting balloon
  Arms: A 1
Device: paclitaxel eluting Taxus stent (Boston Scientific) — paclitaxel-eluting Taxus stents (Boston Scientific) in chronic total occlusion in native coronary arteries
  Arms: A2

SUMMARY:
The aim of the study is to assess the safety and efficacy of a Paclitaxel-eluting PTCA-balloon in combination with bare-metal stenting for treatment of chronic total occlusions in native coronary arteries with reference diameters between 2.5 mm and 4.0 mm.

ELIGIBILITY:
Inclusion Criteria:

* chronic total occlusion
* Thrombolysis in Myocardial Infarction (TIMI) flow 0 or 1
* occlusion in native coronary artery
* indication for percutaneous coronary intervention based on symptoms, prognosis or evidence of ischemia
* reference diameter 2.5 mm to 4.0 mm

Exclusion Criteria:

* saphenous vein graft
* bifurcation lesion with need to stent main and side branch
* left main occlusion
* de-novo stenosis (no occlusion)
* restenosis
* in-stent restenosis
* contraindication for dual antiplatelet therapy with acetylsalicylic acid and clopidogrel for 6 months
* coronary aneurysm at target lesion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Late loss | 6 months

SECONDARY OUTCOMES:
percent diameter stenosis | 6 months
binary angiographic restenosis rate | 6 months
late loss index | 6 months
Target lumen revascularization | 30 days, 6, 12, 24 months
target vessel revascularization | 30 days, 6, 12, 24 months
major adverse cardiac events | 30 days, 6, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Wöhrle, MD; FESC, Principal Investigator — University of Ulm, Ulm, Germany
Locations (2):
- Germany (2):
  - Klinikum Darmstadt, Darmstadt
  - University of Ulm, Ulm

REFERENCES:
- [Background] Wohrle J, Werner GS. Paclitaxel-coated balloon with bare-metal stenting in patients with chronic total occlusions in native coronary arteries. Catheter Cardiovasc Interv. 2013 Apr;81(5):793-9. doi: 10.1002/ccd.24409. Epub 2012 Nov 8. PMID 22511572